CLINICAL TRIAL: NCT06920082
Title: Effects of Progressive Muscle Relaxation Exercises on Sleep, Fatigue and Pain in Pancreatic and Colon Cancer Patients Receiving Chemotherapy
Brief Title: Progressive Muscle Relaxation Exercises on Sleep, Fatigue and Pain in Pancreatic and Colon Cancer Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Sabahattin Zaim University (Other)
Responsible Party: Principal Investigator, Zülfünaz ÖZER, Principal Investigator, Istanbul Sabahattin Zaim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025/01-03
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Cancer; Colon Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive muscle relaxation exercises (Experimental): A total of 18 sessions of progressive relaxation were performed, 3 days a week for 6 weeks
  Interventions: Other: Progressive muscle relaxation exercises
- Control group (No Intervention): Routine maintenance will be applied

INTERVENTIONS:
Other: Progressive muscle relaxation exercises — A total of 18 sessions of progressive relaxation were performed, 3 days a week for 6 weeks.
  Arms: Progressive muscle relaxation exercises

SUMMARY:
With regular practice, relaxation has been found to have many benefits such as reducing sensitivity to pain and fatigue, facilitating the transition to sleep, and improving quality of life. Therefore, this study was planned to examine the effects of progressive muscle relaxation exercises applied to pancreatic and colon cancer patients receiving chemotherapy on sleep, fatigue, and pain.

DETAILED DESCRIPTION:
A total of 18 sessions of progressive relaxation were performed, 3 days a week for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age
* Being able to communicate adequately
* Not having a psychiatric problem
* Those who are determined by a physician to have no physical obstacle to exercise
* Individuals who can use technological devices
* Patients who have had at least 3 cycles

Exclusion Criteria:

* Those with communication problems
* Those with psychiatric problems
* Patients doing any exercise
* Individuals with phones that do not have a voice recording feature
* Individuals with phones that do not have a WhatsApp feature

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-04-07 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | Baseline, pre-intervention (Before progressive muscle relaxation exercises applied)
  The patients were asked to mark their level of pain during relaxation or activities on a 10 cm vertical or horizontal line. In addition, there were forms which were numbered from 1-10 or from 1-100. The number 0 is found at the beginning of the line, and the number 10 is located at the end of the line. A value of 0 shows that there is no pain, and the value 10 expresses unendurable pain. GAS is a common scale in the assessment of pain level. A patient is asked to mark the perceived pain on this line, and the marked point is measured in cm.
Visual Analog Scale | After the intervention (After progressive muscle relaxation exercises applied in week 6)
  The patients were asked to mark their level of pain during relaxation or activities on a 10 cm vertical or horizontal line. In addition, there were forms which were numbered from 1-10 or from 1-100. The number 0 is found at the beginning of the line, and the number 10 is located at the end of the line. A value of 0 shows that there is no pain, and the value 10 expresses unendurable pain. GAS is a common scale in the assessment of pain level. A patient is asked to mark the perceived pain on this line, and the marked point is measured in cm.
The Piper Fatigue Scale | Baseline, pre-intervention (Before progressive muscle relaxation exercises applied)
  It is a 22-item scale that measures four subscales: behavior (6 items), affect (5 items), sensory (5 items), and cognition/mood (6 items). Each item has 11 response categories on a 0-10 metric with verbal descriptors anchoring the endpoints. Each subscale is scored individually and then aggregated together for an overall score, with higher scores reflecting more fatigue.
The Piper Fatigue Scale | After the intervention (After progressive muscle relaxation exercises applied in week 6)
  It is a 22-item scale that measures four subscales: behavior (6 items), affect (5 items), sensory (5 items), and cognition/mood (6 items). Each item has 11 response categories on a 0-10 metric with verbal descriptors anchoring the endpoints. Each subscale is scored individually and then aggregated together for an overall score, with higher scores reflecting more fatigue.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | Baseline, pre-intervention (Before progressive muscle relaxation exercises applied)
  The PSQI is a valid and consistent survey comprising 19 questions to assess the quality and amount of sleep and the existence of a sleep disorder and its level in the previous month. The scale was adapted into the Turkish language by Agargün et al. (1996). The scale consists of seven components that assess patients' subjective sleep quality, sleep delay, use of sleeping medication and dysfunction in daily activities. Each item scores in the range 0-3 points and the total score of the seven components gives the total PSQI score. The total score has a value between 0-21 and a high total score demonstrates a poor quality of sleep. A total PSQI score of ≤5 indicates "good sleep", and a score of>5 indicates "poor sleep"
Pittsburgh Sleep Quality Index (PSQI) | After the intervention (After progressive muscle relaxation exercises applied in week 6)
  The PSQI is a valid and consistent survey comprising 19 questions to assess the quality and amount of sleep and the existence of a sleep disorder and its level in the previous month. The scale was adapted into the Turkish language by Agargün et al. (1996). The scale consists of seven components that assess patients' subjective sleep quality, sleep delay, use of sleeping medication and dysfunction in daily activities. Each item scores in the range 0-3 points and the total score of the seven components gives the total PSQI score. The total score has a value between 0-21 and a high total score demonstrates a poor quality of sleep. A total PSQI score of ≤5 indicates "good sleep", and a score of>5 indicates "poor sleep"

CONTACTS AND LOCATIONS:
Overall Officials: Zülfünaz Özer, PhD, Principal Investigator — İstanbul Sabahattin Zaim Üniversitesi
Locations (1):
- Istanbul Sabahattin Zaim University, Faculty of Health Sciences, Küçükçekmece, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Toraman RL, Eskici Ilgin V. Effect of Virtual Reality Glasses Application on Pain, Anxiety, and Patient Satisfaction During a Transrectal Prostate Biopsy: A Randomized Controlled Trial. Biol Res Nurs. 2024 Oct;26(4):485-497. doi: 10.1177/10998004241236154. Epub 2024 Feb 28. PMID 38418943
- [Result] Loh EW, Shih HF, Lin CK, Huang TW. Effect of progressive muscle relaxation on postoperative pain, fatigue, and vital signs in patients with head and neck cancers: A randomized controlled trial. Patient Educ Couns. 2022 Jul;105(7):2151-2157. doi: 10.1016/j.pec.2021.10.034. Epub 2021 Nov 3. PMID 34785078